CLINICAL TRIAL: NCT07224516
Title: Testing MOUD Scale-Up Strategies in Criminal Legal Settings
Brief Title: Testing MOUD Scale-Up
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-1515; 1UM1DA064515-01 (NIH); Protocol Version 10/10/2025 (Other: UW Madison); SO00004046 (Other: UW Madison); CHESS (Other: UW Madison)
Record Dates: First submitted 2025-10-31; First posted 2025-11-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-10

CONDITIONS: Incarcerated Individuals; Correctional Institutions
Keywords: Correctional staff
MeSH Terms: interventions — United States Substance Abuse and Mental Health Services Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Substance Abuse and Mental Health Services Administration (SAMHSA) Policy Academy (Experimental): Departments of Corrections (DOCs) which previously completed the SAMHSA Policy Academy will be recruited for the Policy Academy.
  Interventions: Behavioral: SAMHSA
- Multi-site Learning Collaborative (LC) (Experimental): The LCs will include learning sessions at baseline and monthly coaching sessions thereafter in the 12 month intervention period to provide training and technical assistance on the study protocol, types of MOUD and their clinical effectiveness, strategies to reduce stigma towards MOUD, approaches to overcoming common MOUD implementation barriers, and strategies to increase use and reduce burden of MOUD.
  Interventions: Behavioral: Learning Collaborative
- Practice as Usual (No Intervention): This arm will conduct practice as usual, not using the updated MOUD practices.

INTERVENTIONS:
Behavioral: SAMHSA — Implement the scale-up of MOUD
  Arms: Substance Abuse and Mental Health Services Administration (SAMHSA) Policy Academy
Behavioral: Learning Collaborative — The LCs will include learning sessions at baseline and monthly coaching sessions thereafter in the 12 month intervention period to provide training and technical assistance on the study protocol, types of MOUD and their clinical effectiveness, strategies to reduce stigma towards MOUD, approaches to overcoming common MOUD implementation barriers, and strategies to increase use and reduce burden of MOUD.
  Arms: Multi-site Learning Collaborative (LC)

SUMMARY:
The goal of this clinical trial is to improve health outcomes for incarcerated individuals by increasing medications for opioid use disorder (MOUD) use, using scalable and cost-effective methods that could be applied more broadly in the criminal justice system.

DETAILED DESCRIPTION:
This trial will evaluate a systems-change approach to scaling medications for opioid use disorder (MOUD) across 120 prisons in 12 U.S. states. Researchers will test two promising, implementation strategies-policy academy and multisite learning collaborative-commonly used in healthcare, education, and community development. The focus on MOUD is driven by strong evidence of its efficacy, low penetration in prisons, significant health inequities among incarcerated populations, and the high risk of overdose deaths during reentry into the community.

ELIGIBILITY:
Inclusion Criteria - Sites:

* Have an interest in embedding or increasing the use of MOUD within their site
* Have the funds to pay for medication for the duration of the study (24 months)
* Agree to implement or continue the use of at least one medication for opioid use disorder
* Have leadership support at all levels including from Secretary of DOC, medical director, wardens, etc.
* Sign a memorandum of Understanding (MOU) or Information Sheet
* Agree to provide data described in the Information Sheet

Exclusion Criteria:

* Failure to meet eligibility criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Reach of systems-change for scaling medications for MOUD | 2 years
  Using the RE-AIM framework, reach is measured by number of MOUD (buprenorphine, methadone, injectable naltrexone) standardized medication units purchased by prisons in a state

SECONDARY OUTCOMES:
Effectiveness of systems-change approach for scaling MOUD | 2 years
  Using the RE-AIM framework, effectiveness is measured by the number of disciplinary infractions and individuals participating in SUD programming
Adoption of systems-change approach for scaling MOUD | 2 years
  Using the RE-AIM framework, adoption is measured as the percentage of prisons that use buprenorphine, methadone, and/or naltrexone
Implementation - IMAT Index | 2 years
  Implementation is measured by Integrating Medications for Addiction Treatment (IMAT) Index (prison level). IMAT is a tool for evaluating and improving how primary care and behavioral health programs integrate MOUD. The scoring ranges from "1-Not Integrated" to "5-Fully Integrated", with intermediate scores of 2 and 4 representing in-between stages. The total IMAT score is calculated by averaging all item scores. This results in a composite rating from 1 to 5, which represents the overall implementation quality.
Implementation - Cascade of Care | 2 years
  Using the RE-AIM framework, implementation is measured by Cascade of Care performance (prison level). Cascade of Care is a framework that tracks progress through different stages of healthcare, from initial contact (like screening or diagnosis) to successful treatment and long-term management. The cascade visualizes how many individuals successfully move from one stage to the next, highlighting points where they are lost from the system.
Implementation - EBI checklist | 2 years
  Using the RE-AIM framework, implementation is measured by Advancing Recovery Framework Implementation of an EBI Checklist (state level). This measure is structured around the Cascade of Care performance (state level), This model helps states assess and improve their treatment systems by tracking individuals' progress from diagnosis through recovery.
Implementation - Partnering | 2 years
  Using the RE-AIM framework, implementation is measured by the level of partnering between DOC and prisons. Measure focuses on the strength and consistency of partnerships between the Department of Corrections (DOC) and individual prisons to support the delivery of evidence-based practices for opioid use disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Molfenter, PhD, Principal Investigator — University of Wisconsin, Madison; Rosemarie Martin, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes